CLINICAL TRIAL: NCT04186767
Title: Significative Weight Loss Impact on Oxidative Stress, Metabolic, Hormonal, Inflammatory and Seminal Parameters of Obese Men.
Brief Title: Weight Loss Impact on Male Fertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Alessandra Renck, Principal Investigator, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 86158918.4.0000.0068
Record Dates: First submitted 2019-04-21; First posted 2019-12-05 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Obesity; Sub Fertility, Male; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Infertility, Male; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Prospective, unicentre, single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weight loss (Experimental)
  Interventions: Dietary Supplement: Very Low Carb Ketogenic Diet

INTERVENTIONS:
Dietary Supplement: Very Low Carb Ketogenic Diet — Patients will be submitted to very low-calorie ketogenic dietary intervention (VLCK) according to the recommendations of the Pronokal® Method program including lifestyle and physical activity guidelines. The ketogenic stage (phase 1-3) consists of a VLCD diet (600-800 kcal / d), with low carbohydrate intake and lipids. The amount of high biological value proteins ranges from 0.8 to 1.2 g / kg of body weight / day. This first stage (ketogenic) is maintained until the patient reaches the goal of reducing the target weight by 80% to be reduced, being variable in time, according to the response of each patient. After this period, it evolved to a non-ketogenic stage, initiating the hypocaloric diet (800 to 1500 Kcal), with progressive introduction of other food groups, reducing weight more slowly. The maintenance stage consists of a balanced diet, ranging from 1500 to 2000 Kcal.

SUMMARY:
This is a prospective non-randomized unicentric clinical trial, characterized by the inclusion of obese (BMI> 35) male with subfertility (sperm count showing low sperm counts and / or motility and / or morphology and / or DNA fragmentation). Patients selected at the endocrinology obesity HC-FMUSP outpatient will be submitted to very low calorie diet (VLCK) for 6 months, being reassessed clinically and laboratorially monthly.

ELIGIBILITY:
Inclusion Criteria:

Obesity in male patients

* Metabolic Syndrome (NCEP-ATP III)
* Alteration of some of the seminal parameters evaluated in conventional seminal analysis

Exclusion Criteria:

* Other causes of hypogonadotrophic hypogonadism

  * Hypergonadotrophic hypogonadism
  * Contraindications for performance of ketogenic diet:
  * Type 1 or type 2 diabetes mellitus in insulin use
  * Food drive
  * Alcoholism or drug addiction
  * Severe psychiatric illness
  * Use of coumarin anticoagulants
  * Hepatic insufficiency
  * Severe renal impairment
  * Hematologic diseases
  * Cancer in activity,
  * Cardiovascular or cerebrovascular diseases (arrhythmias, recent myocardial infarction, unstable angina, decompensated heart failure, recent stroke)
  * Gout
  * Renal or biliary lithiasis
  * Major depression or other serious psychiatric illness.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2023-01-22 (Actual)

PRIMARY OUTCOMES:
Seminal evaluation | Six months
  Spermatic counting will be combined to report
Seminal evaluation | Six months
  Spermatic motility will be combined to report
Seminal evaluation | Six months
  DNA fragmentation will be combined to report

SECONDARY OUTCOMES:
Metabolic response | Six months
  To evaluate the metabolic parameters lipid and glycemic profiles before and after intervention.
Hormonal measurements | Six months
  To evaluate hormonal parameters total testosterone, LH, FSH, insulin before and after intervention.
Inflamatory response | Six months
  To evaluate cytokines TNFa and IL-6 response before and after intervention.
Adipose tissue evaluation | Six months
  To evaluate adipokines: leptin, adiponectin, UCP-1, FGF21, irisin and PGC1a measures before and after intervention.
Microbiota evaluation | Six months
  Evaluate the whole intestinal metagenomics before and after the intervention
Epigenetic evaluation | Six months
  To evaluate the epigenetic methylation profile of spermatozoa before and after the intervention
Body composition changes | Six months
  Apply body composition digital analyser pre and post intervention.
Brow tissue study | Six months
  Thermodynamic evaluation of brown adipose tissue using infrared thermography.
Adipose tissue toxins study | Six months
  Persistent organic pollutants measure: 2,3,7,8- tetrachlorodibenzo-p-dioxin (TCDD)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo, São Paulo, Brazil